CLINICAL TRIAL: NCT06623149
Title: Policy-Induced Conservative Management Prioritization Over Arthroplasty On Knee Osteoarthritis Outcomes
Brief Title: Conservative Management vs. Arthroplasty in Knee Osteoarthritis
Status: Enrolling by invitation | Type: Observational
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Other Study IDs: NOK
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthrosis
Keywords: arthroplasty; exercise; osteoarthritis; weight loss; pain management; quality of ilfe
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Osteoarthritis; Weight Loss; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Old policy: Individuals with knee osteoarthritis referred from a general practitioner to a participating orthopedic department for assessment of eligibility for knee arthroplasty (surgical joint replacement).
  Interventions: Procedure: Current practice
- New policy - non-surgical management: Individuals with knee osteoarthritis referred from a general practitioner to a participating orthopedic department for assessment of eligibility for knee arthroplasty (surgical joint replacement).
  Interventions: Behavioral: Non-Surgical Intervention

INTERVENTIONS:
Behavioral: Non-Surgical Intervention — After referral from the general practitioner to the orthopedic department, the patient is offered a 3-month non-operative treatment program. The conservative program consists of several elements that are offered on an individual basis. The program consists of 3 main elements:
  * Patient education/information
  * Specialized exercise supervised by a physiotherapist
  * Weight loss counseling with a dietician
  Groups: New policy - non-surgical management
Procedure: Current practice — After referral from the general practitioner to the orthopedic department, the patient is assessed by an orthopedic surgeon in the out-patient clinic according to standard practice with a focus on symptoms, history, physical examination, radiography, and an appraisal of the patient's expectations. If an indication for knee arthroplasty is found, the patient is offered knee arthroplasty, and if the patient accepts the offer, he/she is scheduled according to usual practice. If a patient declines the offer, the patient is informed that the hospital cannot offer any additional service, and the patient is referred back to primary care.
  Groups: Old policy

SUMMARY:
The goal of this observational study is to learn about the long-term effects of a non-surgical management programme in people with osteoarthritis that are eligible for a knee joint replacement surgery to treat their knee osteoarthritis (KOA). The main question it aims to answer is:

- Does the non-surgical management programme reduce the proportion of referred patients who are treated with a knee arthroplasty without reducing the health-related quality of life over a two-year perspective?

DETAILED DESCRIPTION:
Knee arthroplasty (joint replacement surgery) is a well-established and effective treatment for knee osteoarthritis (KOA). The incidence of knee arthroplasty has increased in Denmark from 8,000 procedures in 2017 to over 15,000 in 2023, partly due to demographic changes, demands, and the procedures effectiveness. However, concerns remain that some patients undergo surgery without having fully explored non-surgical options.

A growing body of research and public declarations suggest that individuals with KOA may benefit from conservative treatment regimens encompassing physical training, weight loss, and pain management strategies. It is implicitly suggested that surgical procedures may be circumvented or deferred well beyond the span of these conservative measures, without adversely impacting patients' quality of life. Such contentions have garnered the attention of decision-makers in the policy realm.

Consequently, a task force under the Capital Region of Denmark has recently mandated a policy shift requiring public hospitals to establish pathways for conservative, non-operative treatment with a duration of three months that patients must complete prior to considering knee arthroplasty. The aim of this policy alteration is to further prioritize conservative management and curtail the frequency of knee arthroplasty procedures while preserving patients' quality of life. Although the number of surgical procedures could be ostensibly minimized by constraining healthcare service provisions and impeding patient access, the patients' quality of life remains the paramount political objective. Consequently, the task force has decided to assess the impact of the policy change by endorsing and initiating a study to monitor quality, as summarized in the current protocol synopsis.

The new policy is introduced in a step-wise manner at the major hospitals in the Capital Region of Denmark (Copenhagen) from October 1st 2024 to January 1st 2025) and this observational study enrols patients at the hospitals before and after implementation of the new policy to facilitate a comparison of the two policies (new vs old). The enrolled patients are followed for 2 years with regular collection of patient-reported outcomes and medical record reviews.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of knee osteoarthritis.
* Referral from primary care to an orthopedic department at a hospital in The Capital Region of Denmark for treatment of knee osteoarthritis

Exclusion Criteria:

* Referral declined upon initial vetting.
* Not consenting to sharing data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients referred to an orthopedic department at a hospital in The Capital Region of Denmark for treatment of knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients undergoing knee arthroplasty surgery | 2 years
  Percentage of patients who undergo knee replacement surgery in the target joint during the 2-year observation period.
Euroqol 5 dimensions questionnaire (EQ5D) | Average over 2 years (collected at month 0 (enrollment), 3, 6, 9, 12, 18 and 24)
  EQ5D is a standardized patient-reported instrument for use as a measure of health outcome and quality of life. EQ5D is designed for self-completion by respondents and is ideally suited for use in surveys. We will use standard Danish value set to convert the five EQ-5D-5L answers to a single index utility score, and ulti-mately to calculate the QALYs gained by the treatment.

SECONDARY OUTCOMES:
Oxford Knee Score questionnaire | Average over 2 years (collected at month 0 (enrollment), 3, 6, 9, 12, 18 and 24)
  The Oxford Knee Score (OKS) is a 12-item Patient Reported Outcome questionnaire developed specifically to assess the patients perspective on the outcomes of knee arthroplasty with respect to combined pain and physical function. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. Thus, a total score is calculated that ranges from 0 and 48, with 48 indicating the best outcome.
Oxford Knee Score questionnaire | After 2 years (month 24)
  The Oxford Knee Score (OKS) is a 12-item Patient Reported Outcome questionnaire developed specifically to assess the patients perspective on the outcomes of knee arthroplasty with respect to combined pain and physical function. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. Thus, a total score is calculated that ranges from 0 and 48, with 48 indicating the best outcome.
Euroqol 5 dimensions questionnaire (EQ5D) | After 2 years (month 24)
  EQ5D is a standardized patient-reported instrument for use as a measure of health outcome and quality of life. EQ5D is designed for self-completion by respondents and is ideally suited for use in surveys. We will use standard Danish value set to convert the five EQ-5D-5L answers to a single index utility score, and ulti-mately to calculate the QALYs gained by the treatment.
Satisfaction questionnaire | After 1 year (month 12)
  A 5-item questionaire for satisfaction focusing on satisfaction with function of the knee, and the received treatment.
Satisfaction questionnaire | After 2 years (month 24)
  A 5-item questionaire for satisfaction focusing on satisfaction with function of the knee, and the received treatment.
UCLA Physical Activity Scale | Change from baseline after 2 years (month 24)
  The UCLA Activity Scale is a questionnaire used to assess the physical activity levels of patients, particularly those with joint issues, such as knee osteoarthritis or those who have undergone knee arthroplasty. It ranges from 1 to 10, with higher scores indicating higher levels of physical activity. This scale helps clinicians evaluate the functional status of patients and their capacity to perform various physical activities.
UCLA Physical Activity Scale | Change from baseline after 1 year (month 12)
  The UCLA Activity Scale is a questionnaire used to assess the physical activity levels of patients, particularly those with joint issues, such as knee osteoarthritis or those who have undergone knee arthroplasty. It ranges from 1 to 10, with higher scores indicating higher levels of physical activity. This scale helps clinicians evaluate the functional status of patients and their capacity to perform various physical activities.
Copenhagen Knee Range of Motion Scale | After 1 year (month 12)
  The Copenhagen Knee Range of Motion Scale is a clinical tool used to assess and quantify the range of motion in the knee joint. It is particularly useful for evaluating patients with knee osteoarthritis, those undergoing rehabilitation, or those recovering from knee surgeries such as arthroplasty. This scale measures the patient's ability to bend the knee (flexion) and the ability to straighten the knee (extension). The Copenhagen Knee ROM Scale provides a standardized method for healthcare professionals to record knee movement, track progress over time, and guide treatment decisions.
Copenhagen Knee Range of Motion Scale | After 2 years (month 24)
  The Copenhagen Knee Range of Motion Scale is a clinical tool used to assess and quantify the range of motion in the knee joint. It is particularly useful for evaluating patients with knee osteoarthritis, those undergoing rehabilitation, or those recovering from knee surgeries such as arthroplasty. This scale measures the patient's ability to bend the knee (flexion) and the ability to straighten the knee (extension). The Copenhagen Knee ROM Scale provides a standardized method for healthcare professionals to record knee movement, track progress over time, and guide treatment decisions.

OTHER OUTCOMES:
Proportion of patients undergoing knee arthroplasty surgery | 5 years
  Percentage of patients who undergo knee replacement surgery in the target joint over a 5-year observation period.
Costs | During 2 year from enrollment
  Total expenses on healthcare (direct and indirect costs) from enrollment to 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, Professor, Study Chair — The Parker Institute, Bispebjerg Frederiksberg University Hospital, Copenhagen, Denmark; Anders Odgaard, Professor, Study Chair — Rigshospitalet, Denmark
Locations (6):
- Denmark (6):
  - Bispebjerg Frederiksberg Hospital, Copenhagen, Copenhagen
  - Amager Hvidovre Hospital, Copenhagen, Hvidovre
  - Rigshospitalet, Copenhagen
  - herlev Gentofe Hospital, Copenhagen
  - Nordsjællands Hospital, Hillerød
  - Bornholms hospital, Rønne

IPD SHARING:
Plan to Share IPD: Undecided